CLINICAL TRIAL: NCT05801848
Title: Diagnosis of Bone Metabolism in Patients With Inexplicable Lower Back Pain
Status: Active, not recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Rune Toennesen, Md, PhD, Rigshospitalet, Denmark
Other Study IDs: H-19039428
Record Dates: First submitted 2023-03-24; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Lower Back Pain Chronic
Keywords: NaF PET; Bone metabolism; Bone perfusion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic lower back pain patients: Patients with chronic lower back pain where the source could not be identified on MRI scans
  Interventions: Diagnostic Test: [18F]NaF PET/CT scan
- Age matched healthy controls: Healthy individuals without any previously known pain or intervention on lower back
  Interventions: Diagnostic Test: [18F]NaF PET/CT scan

INTERVENTIONS:
Diagnostic Test: [18F]NaF PET/CT scan — Patients will have their lower back scanned using [18F]NaF PET/CT

SUMMARY:
The main goal of this study is to determine if static or dynamic [18F]NaF PET/CT (positron emitting tomography) can identify the source of lower backpain in at least 20% of the patients experiencing lower backpain, yet could not be diagnosed from MRI or CT scans.

DETAILED DESCRIPTION:
Patients with chronic lower backpain are routinely scanned with MR and/or CT to diagnos the source of pain. Larger studies have reported that approximately 20% of patients are given a certain diagnosis from the scans and in the majority of cases the source of the pain is not determined. The use of [18F]NaF PET/CT to map bone perfusion and metabolism is a routine clinical scan that can potentially identify the source of lower backpain in MRI and CT negative patients.

Hypothesis: That [18F]NaF PET/CT bone metabolism and bone perfusion images would contain information that allow the correct diagnosis in at least 20% of patients where MRI and CT images did not reveal pathology.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years
* Chronic lower back pain with no concrete diagnosis after MRI and/or CT
* Under the the care of Rigshospitalets centre for Rheumatology and Spine Disease

Exclusion Criteria:

* previous operation in the lower back area
* Known inflammatory related illness or progressive rheumatism

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with chronic lower back pain where the source could not be identified on MRI scans
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-03-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Abnormal foci of elevated bone metabolism, blood pooling or bone perfusion | 1 hour examination
  [18F]NaF PET/CT scan

CONTACTS AND LOCATIONS:
Overall Officials: Rune Tønnesen, MD PhD, Principal Investigator — Rigshospitalet Centre of Rheumatology and Spine Disease
Locations (1):
- Rigshospitalet - Centre of Rheumatology and Spine Disease, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gamie S, El-Maghraby T. The role of PET/CT in evaluation of Facet and Disc abnormalities in patients with low back pain using (18)F-Fluoride. Nucl Med Rev Cent East Eur. 2008;11(1):17-21. PMID 19173183
- [Result] Kogan F, Broski SM, Yoon D, Gold GE. Applications of PET-MRI in musculoskeletal disease. J Magn Reson Imaging. 2018 Jul;48(1):27-47. doi: 10.1002/jmri.26183. PMID 29969193